CLINICAL TRIAL: NCT06756035
Title: Phase 1a/1b Study of CT-95 in Advanced Cancers Associated With Mesothelin Expression
Brief Title: CT-95 in Advanced Cancers Associated With Mesothelin Expression
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Context Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNTX-CT95-101
Record Dates: First submitted 2024-12-18; First posted 2025-01-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mesothelin-Expressing Tumors; Epithelial Ovarian Cancer; Malignant Pleural Mesothelioma, Advanced; Malignant Peritoneal Mesothelioma, Advanced; Pancreatic Adenocarcinoma Advanced or Metastatic; Lung Adenocarcinoma Metastatic; Cholangiocarcinoma Advanced; Cholangiocarcinoma Non-resectable; Mesothelin-expressing Advanced Cancers; Mesothelin-positive Advanced Malignant Solid Tumors; Colorectal Cancer
Keywords: Phase 1 Dose Escalation Study; CT-95; Advanced, recurrent cancers; Unresectable, metastatic cancers; Cancers associated with mesothelin expression
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Mesothelioma, Malignant; Neoplasm Metastasis; Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CT-95 (Experimental): Each dose cohort will have weekly dosing. Anticipate approximately 8 dose cohorts.
  Interventions: Drug: CT-95

INTERVENTIONS:
Drug: CT-95 — Weekly IV dosing

SUMMARY:
This is a Phase 1a/1b open-label, dose escalation study to evaluate the safety and efficacy of CT-95 (study drug), a humanized T cell engaging bispecific antibody targeting Mesothelin, in subjects with advanced solid tumors associated with Mesothelin expression.

DETAILED DESCRIPTION:
The Phase 1a Dose Escalation portion of the trial will enroll subjects in one of approximately 8 dose escalation cohorts to assess the safety and tolerability of CT-95, as well as determine the maximum tolerated dose (MTD) or other recommended dose(s) for expansion (RDE[s]) for further study in 2 dose optimization cohorts. Subjects will receive CT-95 as a single agent administered once weekly (QW) intravenously (IV) over a 4-week cycle.

The Phase 1b Dose Expansion portion will evaluate CT-95 in indication-specific expansion cohorts

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0 or 1
* Subjects with evaluable disease per RECIST 1.1 or mRECIST
* Subjects with adequate organ function.
* Subjects with advanced cancers associated with mesothelin expression

Exclusion Criteria:

* Uncontrolled significant active infection or any medical or other condition that in opinion of the investigator would preclude the subject's participation in the study.
* Prior treatment with MSLN-targeted CD3 or chimeric antigen receptor T cell (CAR-T) therapy
* Concurrent participation in another investigational clinical trial.
* Evidence of leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Determine the MTD or RD of CT-95 [Safety and Tolerability] | From date of first dose of CT-95 until 28 days following the first dose.
  The frequency of dose-limiting toxicities (DLTs) will be analyzed along with safety and tolerability measures to determine the MTD or RD of CT-95.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From date of first dose of CT-95 for approximately 6 months or until treatment discontinuation, whichever comes first.
  The frequency and severity of adverse events, serious adverse events, and adverse events of special interest will be analyzed.

SECONDARY OUTCOMES:
Evaluate Response Rates [Anti-tumor Activity] | At 8-week intervals from the time of the first dose of CT-95 for approximately 6 months or until treatment discontinuation, whichever comes first
  Overall response rates will be calculated using RECIST 1.1 (and mRECIST for patients with mesothelioma) for CT-95.
Evaluate Progression-free Survival [Anti-tumor Activity] | At 8-week intervals from the time of the first dose of CT-95 for approximately 6 months or until treatment discontinuation, whichever comes first.
  PFS will be summarized using RECIST 1.1 (and mRECIST for patients with mesothelioma) for CT-95.
Evaluate Overall Survival [Survival] | From the time of the first dose of CT-95 until approximately two years post-first dose.
  Overall survival will be summarized for CT-95.
Evaluate the Maximum Serum Concentration (Cmax) [Pharmacokinetics] | From date of first dose of CT-95 for 5 months or until treatment discontinuation, whichever comes first.
  Serum concentrations of CT-95 analyzed as a function of time relative to dosing will be calculated.
Evaluate the Area Under the Curve (AUC) [Pharmacokinetics] | From date of first dose of CT-95 for 5 months or treatment discontinuation, whichever comes first.
  The AUC of CT-95 analyzed as a function of time relative to dosing will be calculated.
Evaluate Anti-Drug Antibodies [Immunogenicity] | From date of first dose of CT-95 for 5 months or until treatment discontinuation, whichever comes first.
  Incidence and titer of ADAs will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chagin, MD, Study Director — Context Therapeutics Inc.
Locations (7):
- United States (7):
  - Context Investigational Site, Denver, Colorado
  - Context Investigational Site, Chicago, Illinois
  - Context Investigational Site, Grand Rapids, Michigan
  - Context Investigational Site, Hackensack, New Jersey
  - Context Investigational Site, Philadelphia, Pennsylvania
  - Context Investigational Site, Nashville, Tennessee
  - Context Investigational Site, San Antonio, Texas